CLINICAL TRIAL: NCT02303444
Title: RIFTOS MKI - Radioactive Iodine reFractory Asymptomatic Patients in Differentiated Thyroid Cancer - an Observational Study to Assess the Use of Multikinase Inhibitors
Brief Title: An Observational Study in Differentiated Thyroid Cancer Which is Radioactive Iodine (RAI) Refractory to Assess the Use of Multikinase Inhibitors
Acronym: RIFTOS MKI
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17852; NX1401 (Other: Company internal)
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Thyroid Neoplasms
Keywords: Progressive radioactive iodine refractory differentiated thyroid carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MKI patients: Asymptomatic patients with RAI-refractory progressive DTC for whom there is a decision to initiate MKIs at study entry. For patients on sorafenib, treatment start and stop dates will be collected along with any adverse events observed.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Other Multikinase inhibitors
- non-MKI patients: Asymptomatic patients with RAI-refractory progressive DTC for whom there is a decision to not initiate MKIs at study entry. For patients on sorafenib, treatment start and stop dates will be collected along with any adverse events observed.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Other Multikinase inhibitors

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients can get sorafenib at any time during study.
Drug: Other Multikinase inhibitors — Patients can get MKIs at any time during study.

SUMMARY:
The purpose of the study was to assess the use of Multikinase Inhibitors (MKIs) in the treatment of patients with a progressive differentiated thyroid carcinoma (DTC) refractory to radioactive iodine (RAI) who do not have any symptoms.

DETAILED DESCRIPTION:
The primary objective of this study was to compare time to symptomatic progression (TTSP) from study entry in asymptomatic patients with RAI-refractory progressive DTC for whom there is a decision to initiate MKIs at study entry with that of asymptomatic patients with RAI-refractory progressive DTC for whom there is a decision to not initiate MKIs at study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically documented DTC (papillary, follicular, Hurthle cell, and poorly differentiated carcinoma)
* DTC refractory to RAI
* Radiological progression and preferably according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* No symptoms due to DTC
* >/=1cm diameter of lesion confirmed by radiological exam
* Life expectancy of at least 6 months

Exclusion Criteria:

* Plan to be treated according to a clinical trial protocol for intervention including a locoregional therapy or systemic therapy
* Previous treatment with MKIs for advanced disease
* Hospice patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any setting that provides treatment for progressive asymptomatic RAI refractory DTC
Sampling Method: Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Time to symptomatic progression (TTSP) from study entry | Up to 6 years
  TTSP is defined as the time interval from the day of study entry to the date of first symptomatic progression. Patients who do not have a symptomatic progression at the time of analysis will be censored at the date of their last evaluable assessment.

SECONDARY OUTCOMES:
Overall survival (OS) from time of study entry | Up to 6 years
  Defined as the time interval from the date of study entry to death due to any cause. Patients alive at the time of analysis will be censored at the last date known to be alive.
Progression free survival (PFS) from time of study entry | Up to 6 years
  Defined as the time interval from the date of study entry to date of first progression or death due to any cause, whichever comes first. The actual date of tumor assessments will be used for this calculation. Patients without a progression or death will be censored at their last evaluable date of tumor evaluation.
OS from time of being diagnosed as radioactive iodine (RAI) refractory | Up to 6 years
  Defined as the time interval from the day of being diagnosed as RAI refractory to death due to any cause. Patients alive at the time of analysis will be censored at the last date known to be alive.
Post-progression survival (PPS) from time of symptomatic progression | Up to 6 years
  Defined as the time interval from the date of symptomatic progression to death due to any cause. Patients without symptomatic progression will be excluded from analysis and patients who are alive at the time of analysis will be censored at the last date when they were known to be alive.
OS from initiation of the first Multikinase Inhibitor (MKI) | Up to 6 years
  Defined as the time interval from the day of start of the first MKI to death due to any cause. Patients alive at the time of analysis will be censored at the last date when they were known to be alive.
PFS from initiation of first MKI | Up to 6 years
  Defined as the time interval from the day of start of first MKI to date of first progression or death due to any cause, whichever comes first. The actual date of tumor assessments will be used for this calculation. Patients without a progression or death will be censored at their last evaluable date of tumor evaluation.
OS from initiation of any systemic treatment regimen | Up to 6 years
  Defined as the time interval from the date of start of any systemic treatment regimen to death due to any cause. Patients alive at the time of analysis will be censored at the last date known to be alive.
PFS from initiation of any systemic treatment regimen | Up to 6 years
  Defined as the time interval from the date of start of any systemic treatment regimen to date of first progression or death due to any cause, whichever comes first. Patients without a progression or death will be censored at their last evaluable date of tumor evaluation.
Duration of each systemic treatment regimen | Up to 6 years
  Defined as the time interval from the day of start of a treatment to the date of permanent discontinuation of a treatment (regardless of the reason for discontinuation including death). It includes interruption or drug holiday.
Response assessment to each systemic treatment regimen according to the categories "Complete Response", "Partial Response", "Stable Disease", "Clinical Progression", "Radiological Progression", and "Not evaluable at this visit" | Up to 6 years
  In case of "Clinical Progression" the CRF will ask for the presence of specific symptoms.
OS from initiation of sorafenib | Up to 6 years
  Defined as the time interval from the day of start of sorafenib to death due to any cause. Patients alive at the time of analysis will be censored at the last date known to be alive.
PFS from initiation of sorafenib | Up to 6 years
  Defined as the time interval from the date of start of sorafenib to date of first progression or death due to any cause, whichever comes first. Patients without a progression or death will be censored at their last evaluable date of tumor evaluation.
Daily dose of sorafenib per patient throughout the treatment period | Up to 6 years
Number of adverse events during treatment with sorafenib | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (34):
- United States (16):
  - Birmingham, Alabama
  - Los Angeles, California
  - Torrance, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Plantation, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - The Bronx, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Dallas, Texas
- Multiple Locations, Algeria
- Multiple Locations, Argentina
- Multiple Locations, Brazil
- Multiple Locations, Egypt
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Greece
- Multiple Locations, India
- Multiple Locations, Japan
- Multiple Locations, Lebanon
- Multiple Locations, Mexico
- Multiple Locations, Netherlands
- Multiple Locations, Philippines
- Multiple Locations, Russia
- Multiple Locations, Saudi Arabia
- Multiple Locations, Spain
- Multiple Locations, Taiwan
- Multiple Locations, Turkey (Türkiye)

REFERENCES:
- [Derived] Gianoukakis AG, Choe JH, Bowles DW, Brose MS, Wirth LJ, Owonikoko T, Babajanyan S, Worden FP. Real-world practice patterns and outcomes for RAI-refractory differentiated thyroid cancer. Eur Thyroid J. 2024 Jan 24;13(1):e230039. doi: 10.1530/ETJ-23-0039. Print 2024 Feb 1. PMID 38096102
- [Derived] Brose MS, Smit JWA, Lin CC, Tori M, Bowles DW, Worden F, Shen DH, Huang SM, Tsai HJ, Alevizaki M, Peeters RP, Takahashi S, Rumyantsev P, Guan R, Babajanyan S, Ozgurdal K, Sugitani I, Pitoia F, Lamartina L. Multikinase Inhibitors for the Treatment of Asymptomatic Radioactive Iodine-Refractory Differentiated Thyroid Cancer: Global Noninterventional Study (RIFTOS MKI). Thyroid. 2022 Sep;32(9):1059-1068. doi: 10.1089/thy.2022.0061. PMID 35950621
- [Derived] Porcelli T, Luongo C, Sessa F, Klain M, Masone S, Troncone G, Bellevicine C, Schlumberger M, Salvatore D. Long-term management of lenvatinib-treated thyroid cancer patients: a real-life experience at a single institution. Endocrine. 2021 Aug;73(2):358-366. doi: 10.1007/s12020-021-02634-z. Epub 2021 Feb 3. PMID 33537956
- [Derived] Brose MS, Smit J, Lin CC, Pitoia F, Fellous M, DeSanctis Y, Schlumberger M, Tori M, Sugitani I. Timing of multikinase inhibitor initiation in differentiated thyroid cancer. Endocr Relat Cancer. 2017 May;24(5):237-242. doi: 10.1530/ERC-17-0016. Epub 2017 Mar 7. PMID 28270435